CLINICAL TRIAL: NCT03127137
Title: Do Cervical Interlaminar Epidural Steroid Injections With Low-dose Lidocaine Cause Transient Objective Upper Extremity Weakness? A Prospective Randomized Controlled Trial
Brief Title: CESI With Low Dose Lidocaine and Transient Weakness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00204980
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Cervical Radiculitis; Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial using control arm plus 2 arm experimental (placebo and active drug)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be blinded to group assignment. Outcome assessor will also be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group 1 (Active Comparator): Experimental Group 1 will receive Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL 1% lidocaine (total volume 4 cc)
  Interventions: Drug: Experimental Group 1 triamcinolone and lidocaine
- Experimental Group 2 (Placebo Comparator): Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL preservative saline (total volume 4 cc)
  Interventions: Drug: Experimental Group 2 triamcinolone and saline

INTERVENTIONS:
Drug: Experimental Group 1 triamcinolone and lidocaine — Experimental Group 1 will receive Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL 1% lidocaine (total volume 4 cc)
  Other Names: Experimental Group 1
  Arms: Experimental Group 1
Drug: Experimental Group 2 triamcinolone and saline — Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL preservative saline (total volume 4 cc)
  Other Names: Experimental Group 2
  Arms: Experimental Group 2

SUMMARY:
Cervical radicular pain is relatively common, often treated with epidural steroid injection (ESI), when conservative treatments like oral analgesics, physical therapy and activity modification have failed. There are no universal clinical practice guidelines for the use of diluents when CESI are performed.

Interlaminar CESI may be performed with or without the use of local anesthetics, due to training bias or theoretical concerns of weakness. CESI without the benefit of local anesthetic as a steroid diluent increases the latency of pain relief and may decrease diagnostic information immediately after a CESI with regard to pain generators responsible for symptoms, and may potentially decrease patient satisfaction.

By evaluating the effects of local anesthetic as a diluent during interlaminar cervical ESI, we will enhance the safety of this treatment with regard to expectations of objective motor weakness as well as post procedure pain control and patient satisfaction in the recovery phase after the injection procedure.

Research Question:

Does lidocaine versus saline as a steroid diluent effect objective upper extremity strength following cervical epidural steroid injection in patients being treated for cervical radiculitis?

Null Hypothesis:

Cervical epidural steroid injections that include local anesthetic as a diluent have no effect on objective upper extremity strength following the injection.

We hypothesized that cervical epidural lidocaine will cause an objective decrease in strength in functional movements of the upper extremity.

DETAILED DESCRIPTION:
Experimental Groups: Prospective, randomized, controlled, double blinded trial in patients undergoing CESI for symptoms of cervical radiculitis.

Group #1: Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL 1% lidocaine (total volume 4 cc).

Group #2: Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL preservative saline (total volume 4 cc).

Adults who are eligible to have a CESI with triamcinolone for treatment of cervical radiculitis at the Northwestern Anesthesiology Pain Medicine Center will be approached by authorized research personnel prior to a patient's CESI is performed and will obtain informed consent from patients who agree to participate.

In every subject (Group 1 and Group 2) a pre-procedure NRS pain score, and presence of subjective or objective symptoms of UE weakness will be recorded. Bilateral handgrip, wrist extension, elbow flexion, and elbow extension strength (myotomes C5-T1) will be measured by a trained research assistant prior to the injection procedure using a handheld JAMAR® PLUS+ digital dynamometer (Sammons Preston, Bollingbrook, IL) for hand grip strength and a push/pull handheld hydraulic dynamometer (Balego and Associates Inc., St. Paul, MN) for arm strength assessment. Three baseline strength measurements will be recorded for each strength test. Measurements will be taken prior to and 30 minutes following the injection procedure. Patients in Group #1 and Group #2 will also be queried with the Upper Extremity Functional Index (UEFI) before the injection procedure and again 1 day after the procedure (administered via telephone).

For Group 1 and Group 2, patients will be randomized to treatment group based on a random computer-generated schedule. Participants will be blinded to the group to which they are randomized. All standard procedures for CESIs will be followed as is standard practice including time out, skin prep, hemodynamic monitoring, image guidance etc.

Per randomization, triamcinolone acetonide 80 mg (Kenalog) (E. R. Squibb & Sons Limited, Uxbridge UK) will be combined with 2mL Lidocaine 1% or 2 mL preservative free saline and will be injected during the CESI procedure. In all cases, the total injectate volume will be 4 mL in all cases. All injections will be image guided with fluoroscopy, as is the current standard practice. Fluoroscopy time will be recorded.

The participant will be discharged from the clinic with written discharge instructions (current standard practice).

Participants will be telephoned by clinic personnel 1 day after the CESI to assess for subjective weakness in the hands or arms as well as any other adverse reactions. As above, the Upper Extremity Functional Index will be administered at this time.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 18 years or older who will undergo CESI for treatment of cervical radiculitis

Exclusion Criteria:

* Patient refusal
* Lack of consent
* Any contraindication to CESI
* Inability to communicate with staff or to participate in follow up
* Inability to perform handgrip or arm strength testing
* Cervical spinal cord lesions
* Cerebrovascular, demyelinating or other neuromuscular muscular disease
* Patient request for or requirement of conscious sedation for the injection procedure
* Pregnancy
* Breast feeding
* Sensitivity to amides
* History of allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peloso P, Gross A, Haines T, Trinh K, Goldsmith CH, Burnie S; Cervical Overview Group. Medicinal and injection therapies for mechanical neck disorders. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD000319. doi: 10.1002/14651858.CD000319.pub4. PMID 17636629
- [Background] Stav A, Ovadia L, Sternberg A, Kaadan M, Weksler N. Cervical epidural steroid injection for cervicobrachialgia. Acta Anaesthesiol Scand. 1993 Aug;37(6):562-6. doi: 10.1111/j.1399-6576.1993.tb03765.x. PMID 8213020
- [Background] Cicala RS, Thoni K, Angel JJ. Long-term results of cervical epidural steroid injections. Clin J Pain. 1989 Jun;5(2):143-5. doi: 10.1097/00002508-198906000-00003. PMID 2520395
- [Background] Botwin KP, Castellanos R, Rao S, Hanna AF, Torres-Ramos FM, Gruber RD, Bouchlas CG, Fuoco GS. Complications of fluoroscopically guided interlaminar cervical epidural injections. Arch Phys Med Rehabil. 2003 May;84(5):627-33. doi: 10.1016/s0003-9993(02)04862-1. PMID 12736872
- [Background] Rowlingson JC, Kirschenbaum LP. Epidural analgesic techniques in the management of cervical pain. Anesth Analg. 1986 Sep;65(9):938-42. PMID 3017152
- [Derived] McCormick ZL, Burnham T, Cunningham S, Kendall RW, Bougie D, Teramoto M, Walega DR. Effect of low-dose lidocaine on objective upper extremity strength and immediate pain relief following cervical interlaminar epidural injections: a double-blinded randomized controlled trial. Reg Anesth Pain Med. 2020 Oct;45(10):767-773. doi: 10.1136/rapm-2020-101598. Epub 2020 Aug 11. PMID 32784231

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 159 subjects were assessed for eligibility. 27 declined to participate. 2 could not perform pre-study strength testing. 7 requested sedation for the injection.
Period: Overall Study
Arm/Group | Experimental Group 1 | Experimental Group 2
Started | 62 | 61
Completed | 60 | 60
Not Completed | 2 | 1
Not completed — Requested sedation after consent | 1 | 0
Not completed — Malfunction in electronic data collection | 1 | 0
Not completed — Post procedure testing could not be obtained | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group 1 With Lidocaine: Experimental Group 1 will receive Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL 1% lidocaine (total volume 4 cc)
  Experimental Group 1 triamcinolone and lidocaine: Experimental Group 1 will receive Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL 1% lidocaine (total volume 4 cc)
- Experimental Group 2 With Saline: Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL preservative saline (total volume 4 cc)
  Experimental Group 2 triamcinolone and saline: Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL preservative saline (total volume 4 cc)
- Total: Total of all reporting groups
Arm/Group | Experimental Group 1 With Lidocaine | Experimental Group 2 With Saline | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years]
  Years | 56.6 (14) | 56.3 (13.4) | 56.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 30 | 34 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: BMI (kg/m^2)] | 26.5 (4.9) | 29.2 (6.1) | 27.8 (5.5)
Number of Participants with radicular pain based on myotome location [Count of Participants; unit: Participants] — Radicular pain based on the location of the myotome determined by the physician. (grouping of muscles controlled by a single nerve).
  Participants
    c 5 myotome | 15 | 13 | 28
    c 6 myotome | 29 | 30 | 59
    c 7 myotome | 12 | 9 | 21
    c 8 myotome | 0 | 1 | 1
    Missing myotome location | 4 | 7 | 11
Numerical rating score(NRS) for pain [Mean (Standard Deviation); unit: score on a scale] — NRS is an 11 point pain scale where 0 is no pain (good) and 10 is worst pain imaginable (poor)
  score on a scale | 4.9 (2.3) | 5.4 (2.4) | 5.2 (2.3)
Number of participants with unilateral or bilateral symptoms [Number; unit: participants] — Laterally of the symptoms in percent frequency. Unilateral (one sided) or bilateral (both side) before treatment .
  participants
    Unilateral | 47 | 47 | 94
    Bilateral | 13 | 11 | 24
    Missing | 1 | 1 | 2
Physical exam- weakness in any myotome, freq (%) [Number; unit: participants]
  Yes weakness | 3 | 12 | 15
  No weakness | 54 | 47 | 101
  Missing data | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Strength in Both Groups After CESI.
Description: Change in strength in both groups greater than or equal to 20% weakness in one or more myotomes 30 minutes after CESI using a hand held Dynamometer.
Time Frame: 30 minutes after the CESI procedure
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Group 1 With Lidocaine: Experimental Group 1 triamcinolone and lidocaine: Experimental Group 1 will receive Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL 1% lidocaine (total volume 4 cc)
- Experimental Group 2 With Saline: Experimental Group 2 triamcinolone and saline: Interlaminar cervical ESI at the C7-T1 level with triamcinolone 80 mg + 2 mL preservative saline (total volume 4 cc)
Arm/Group | Experimental Group 1 With Lidocaine | Experimental Group 2 With Saline
Number analyzed (Participants) | 60 | 60
Participants
  Yes, greater or equal to 20% weakness in greater or equal to 1 or more myotome | 25 | 30
  No, greater or equal to 20% weakness in greater or equal to 1 or more myotome | 35 | 30
Statistical Analysis 1: Comparison: Experimental Group 1 With Lidocaine vs Experimental Group 2 With Saline; Test type: Superiority; p = .05, Fisher Exact — The reported p-value was calculated

2. Secondary Outcome: Number of Participants With Pain Reduction Post Procedure
Description: A greater than or equal to 50% reduction in change in average pain score before and after the CESI procedure.
Time Frame: 30 minutes after the CESI procedure.
Population: Patients whose baseline and post-NRS scores were both zero were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1 With Lidocaine | Experimental Group 2 With Saline
Number analyzed (Participants) | 59 | 57
Participants
  Experienced greater than or equal to 50% reduction in pain | 19 | 12
  Less than 50% reduction in pain | 40 | 45
Statistical Analysis 1: Comparison: Experimental Group 1 With Lidocaine vs Experimental Group 2 With Saline; Test type: Superiority; Risk Ratio (RR) = 1.53, 95% CI 2-sided [.82 to 2.86]

ADVERSE EVENTS:
Time Frame: 24 hours after the procedure.
Arm/Group | Experimental Group 1 With Lidocaine | Experimental Group 2 With Saline
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 6/60 | 7/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group 1 With Lidocaine (N=60) | Experimental Group 2 With Saline (N=60)
Vasovagal (Nervous system disorders) | 1 (1) | 2 (2) — Vasovagal response
Cardiac rhythm changes (Cardiac disorders) | 2 (2) | 0 (0) — Change in heart rate patern
Pain at injection site (Nervous system disorders) | 1 (1) | 1 (1) — Pain at the injection site where the needle was placed.
Paraesthesia/numbness (Nervous system disorders) | 2 (2) | 4 (4) — Numbness in the hands after the procedure.

LIMITATIONS AND CAVEATS:
Post procedural strength was not assessed beyond 30 minutes. Pain and pain-related outcomes are subjective and variable. It may have been beneficial to have a global impression of change (PGIC)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT03127137/Prot_SAP_001.pdf